CLINICAL TRIAL: NCT04376567
Title: Understanding the Patient-Centered Outcomes for One-stage and Two-stage Brachial Basilic Upper Extremity Arteriovenous Fistulas: A Pilot Trial
Brief Title: Outcomes for One-stage and Two-stage Brachial Basilic Arteriovenous Fistulas
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI is leaving the institution and the trial will be not resuming.
Sponsor: Tze-Woei Tan (Other)
Collaborators: University of Utah (Other); Rancho Los Amigos National Rehabilitation Center (Other)
Responsible Party: Sponsor-Investigator, Tze-Woei Tan, Clinical Associate Professor of Surgery, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0702
Record Dates: First submitted 2020-01-15; First posted 2020-05-06 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: End Stage Renal Failure; Hemodialysis Access Failure; Arterio-venous Fistula
Keywords: Renal failure; Upper extremity arteriovenous fistula; Brachial basilic arteriovenous fistula
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Assigned to either a one-stage or two-stage approach for brachial-basilic arteriovenous fistula (BBAVF) creation in a 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One stage approach (Active Comparator): To create a brachial-basilic arteriovenous fistula (BBAVF) using a one-stage approach. The arteriovenous anastomosis is performed and the basilic vein is transposed during the same procedure.
  Interventions: Procedure: One stage approach
- Two Stage approach (Active Comparator): To create a BBAVF using a two-stage approach, the arteriovenous anastomosis is performed during the first procedure. The superficialization or transposition of the fistula is then performed 6 to 8 weeks later, after the fistula has matured.
  Interventions: Procedure: One stage approach

INTERVENTIONS:
Procedure: One stage approach — Upper extremity brachial basilic arteriovenous fistula will be created either using one stage or two stage approach.
  Other Names: Two stage approach

SUMMARY:
An arteriovenous (AV) fistula is essential for patients with kidney failure on dialysis. There is no clear data on the best method to create a new brachial basilic AV fistula (BBAVF), so the choice between a single procedure and two separate procedures is left to the surgeon. Both approaches are standard care. This study aims to compare patient-centered outcomes and quality of life by randomly assigning patients needing a BBAVF to either a one-stage or two-stage procedure.

DETAILED DESCRIPTION:
The aim of the pilot trial is to compare the outcomes of patients with end stage kidney failure (ESKD) who are candidates for a new brachial basilic arteriovenous fistula (BBAVF). Patients will be randomized to either one-stage or two-stage BBAVF procedure, both standard of care for creating BBAVF. The main outcome will be primary clinical functional patency, defined as successful use of BBAVF over a continuous 4-week period without any need for additional procedure on the BBAVF. The secondary outcomes are fistula-related complications, duration of central venous catheter (CVC) for those on dialysis, and quality of life (QoL) measures. The study hypothesizes that the primary patency will be superior following the two-stage BBAVF procedure compare to one-stage procedure. However, CVC-related complications are expected to be higher following the two-stage procedure compared to the one-stage procedure. Patient will be followed for a minimum duration of 12-months per subject.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. ESRD receiving hemodialysis in need for new hemodialysis access;
3. Candidate for one-stage and two-stage BVT procedure as judged by the enrolling investigator;
4. Greater than 3 mm diameter of upper arm basilic vein on venous duplex scan;
5. Life expectancy ≥ 12 months;

Exclusion Criteria:

1. Life expectancy < 12 months;
2. Brachial artery stenosis or occlusion;
3. A documented hypercoagulable state (defined as a known blood disorder associated with venous or arterial thrombosis);
4. Current immunosuppressive medication, chemotherapy or radiation therapy;
5. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tze-Woei Tan, MD, Principal Investigator — Banner University Medical Center Tucson/University of Arizona
Locations (1):
- Banner University Medical Center Tucson, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | One Stage Approach | Two Stage Approach
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | One Stage Approach | Two Stage Approach | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Dialysis [Count of Participants; unit: Participants] | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Successful Use of Arteriovenous Fistula for Dialysis
Description: Functional clinical patency means the number of participants who were able to use their brachial basilic arteriovenous fistula (BBAVF) successfully for dialysis within 6 months of surgical creation. It refers to using two dialysis needles in at least 75% of dialysis sessions over four weeks without need for additional procedure or surgery, as determined by their providers.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | One Stage Approach | Two Stage Approach
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

2. Secondary Outcome: Number of Participants Who Had Catheter Related Complications
Description: Number of participants with dialysis catheter related complications, including infection, procedure to exchange catheter due to malfunction.
  outcomes of Primary Clinical Functional Patency or CVC-related bacteremia or death
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | One Stage Approach | Two Stage Approach
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

3. Secondary Outcome: Number of Participants Who Had > 3 Months of Catheter Dependency After Arteriovenous Creation
Description: Number of participants who had > 3 months of catheter dependency after arteriovenous fistula creation
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | One Stage Approach | Two Stage Approach
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

4. Secondary Outcome: Patient-Reported Outcomes Measurement Information System Scores Over 6 Months
Description: Average quality of life scores assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) for physical function, fatigue, sleep disturbance, and ability to participate in social roles and activities. Data are presented as T-score, which are standardized scores with a mean of 50 and a standard deviation for the reference population (typically the US general population). A T-score of 50 represents the population average. A higher T-score indicates more of the concept being measured and lower T-score indicate less.
Time Frame: 6-month
Population: Participate did not complete PROMIS questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | One Stage Approach | Two Stage Approach
Number analyzed (Participants) | 1 | 0
score on a scale
  Physical function (T-score) | 37.5 (33.2) |
  Fatigue (T-score) | 52.3 (61.6) |
  Sleep disturbance (T-score) | 53.6 (39.6) |
  Ability to participate in social roles and activities (T-score) | 44.7 (23.7) |

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | One Stage Approach | Two Stage Approach
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Study was terminated early due to low enrollment and PI leaving the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT04376567/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT04376567/ICF_001.pdf